CLINICAL TRIAL: NCT07062185
Title: An Open-label, Single-arm, Single-center Study Evaluating the Safety, Pharmacokinetics, and Preliminary Efficacy of ENC1018 Capsules in Patients With Moderate-to-severe Active Ulcerative Colitis (UC)
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of ENC1018 Capsules in Patients With Moderate-to-severe Active Ulcerative Colitis (UC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, wang xin, Pofessor, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENC1018-UC-01
Record Dates: First submitted 2025-03-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC)
Keywords: ENC1018; moderate to severe active Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ENC1018 capsule administration group (Experimental)
  Interventions: Drug: ENC1018 capsule administration group

INTERVENTIONS:
Drug: ENC1018 capsule administration group — ENC1018 capsules were taken orally once a day for 14 days.

SUMMARY:
This is an open-label, single-arm, single-center study to evaluate the safety, pharmacokinetics, and efficacy signal of ENC1018 capsules in patients with moderate-to-severe active ulcerative colitis (UC).

DETAILED DESCRIPTION:
The study will enroll about 10 diagnosed patients with moderate-to-severe active UC. Each patient will receive an oral dose of ENC1018 capsules once daily for 14 consecutive days after enrollment. Before each dose, patients must fast for at least 2 hours to remain in a fasting state, and no food should be consumed for at least 2 hours after dosing. The entire study period includes a screening phase of up to 3 weeks, a 14-day treatment period, and a 2-week follow-up period. The total duration of the trial is up to 49 days, and patients will be hospitalized during the treatment period. Blood and fecal samples will be collected during the study for PK evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years, male or female.
2. Ulcerative colitis has been diagnosed at least 3 months before screening, and the diagnosis must be confirmed by endoscopy or radiology and histology.
3. Have moderate to severe active ulcerative colitis, defined as a modified Mayo score ≥6.
4. Poor response or intolerance to at least one conventional therapy (aminosalicylic acids, corticosteroids, or immunomodulators) or biologics (anti-TNF, anti-α4β7 integrin, or anti-IL-12/23 antibody drugs) as determined by the investigator.
5. If subjects are taking oral aminosalicylic acids or oral glucocorticoids, their doses must remain stable for at least 2 weeks prior to enrollment and for the duration of the study.
6. Voluntarily sign the informed consent and be willing to follow the research procedures and complete the test in accordance with the protocol.

Exclusion Criteria:

1. Diagnosed with undefined colitis, infectious colitis, ischemic colitis, fulminant colitis, toxic megacolon, or other chronic intestinal diseases other than UC such as Crohn's disease (CD), intestinal tuberculosis, radiation enteritis, and intestinal belcet's disease.
2. Never received any previous treatment for UC.
3. Participated in any other clinical trial within 3 months prior to screening (except those who have only participated in clinical trial screening without using the experimental drug).
4. Subjects with a history of alcohol or drug abuse and complete abstinence for less than 6 months before enrollment.
5. Received any live vaccine within 6 weeks prior to enrollment or planned to receive any live vaccine during the study period or within 6 weeks after the last use of the investigational drug.
6. Experienced major trauma or major surgery within 4 weeks before enrollment;
7. Have any other gastrointestinal diseases that may affect the absorption of oral drugs or have undergone gastrectomy or gastric bypass surgery.
8. Assessed by investigator as needing or receiving total parenteral nutrition and/or total enteral nutrition.
9. Allergy to the test drug or its ingredients.
10. Surgical treatment for ulcerative colitis, including but not limited to ostomy, ileal pocket anal anastomosis, and intestinal resection, is required during prior or anticipated study.
11. Pregnant and lactating women; Or women of childbearing age who have positive blood pregnancy test results during screening; Or had a birth plan throughout the trial period and within 3 months after the end of the study; Or unwilling to use one or more types of physical contraception during the trial and for three months after the end of the study.
12. The investigator believes that participation in this study is not appropriate for other reasons; Or other conditions that may confuse or interfere with the safety, tolerability, or pharmacokinetic evaluation of the investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) and Serious Adverse Events (SAE); | Day 1 - Day 28
Tmax of ENC1018 and its major metabolites in patients with moderate-to-severe active ulcerative colitis (UC). | Day 1 - Day 17
Cmax of ENC1018 and its major metabolites in patients with moderate-to-severe active ulcerative colitis (UC). | Day 1 - Day 17
AUC of ENC1018 and its major metabolites in patients with moderate-to-severe active ulcerative colitis (UC). | Day 1 - Day 17

SECONDARY OUTCOMES:
Fecal PK parameters of ENC1018 and its major metabolites: cumulative excretion amount (Ae); | Day 1- Day 17
Changes in partial Mayo scores (excluding endoscopy scores from the complete modified Mayo score) from baseline; | Day 1- Day 28
Changes in the pharmacodynamic biomarker hsCRP and fecal calcarein from baseline. | Day 1- Day 28
Fecal PK parameters of ENC1018 and its major metabolites: excretion fraction (Fe); | Day 1- Day 17
Changes in defecation frequency (SF) scores from baseline; | Day 1- Day 28
Changes in blood in the stool (RB) scores from baseline; | Day 1- Day 28

IPD SHARING:
Plan to Share IPD: No